CLINICAL TRIAL: NCT05832671
Title: Ultrasound Guided Erector Spinae Muscle Block on Postoperative Pain in Pediatric Patient Undergoing Hip Reconstruction Surgeries
Brief Title: Ultrasound Guided Erector Spinae Muscle Block in Pediatric Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Abbas Hassan, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP54361
Record Dates: First submitted 2023-03-31; First posted 2023-04-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Hip Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US guided erector spinae muscle block (Active Comparator): patients will receive US-guided erector spinae muscle block with a total volume of 0.4 mg/kg of 0.25% bupivacaine.
  Interventions: Procedure: Erector Spinae muscle block
- ultrasound-guided caudal block (Active Comparator): patients will receive an ultrasound-guided caudal block with 2.5 mg/kg of 0.25% bupivacaine to be injected over one minute period while observing an ultrasound longitudinal image.
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: Erector Spinae muscle block — In the ESB group, the patient will be placed in the lateral position. The site of surgery is upward. After skin preparation using 10% povidone-iodine, a high-frequency linear ultrasound transducer will be placed over the ipsilateral site of surgery 1-2 cm lateral to the spine at the T10 level, counting upward from the sacrum. After identifying the erector spinae muscles and transverse process, a needle will be inserted with an in-plane technique in the craniocaudal direction
  Arms: US guided erector spinae muscle block
Procedure: caudal block — In the CB group, patients will be placed in a lateral position. An ultrasound transducer is first placed transversely at the midline to obtain a transverse view of the 2 cornua, the sacrococcygeal ligament, sacral bone, and sacral hiatus. At this position, the ultrasound transducer will be twisted to 90° to obtain longitudinal views of the sacrococcygeal ligament and sacral hiatus and will be subsequently placed between the 2 cornua and on visualization of the frog sign (the 2 sacral cornua identified as 2 hyperechoic reverse U-shaped structure) the needle will be inserted into the sacral canal under direct real-time longitudinal visualization. After negative aspiration for blood or cerebrospinal fluid, bupivacaine (0.25%) 2.5 mg/kg will be injected over a one minute period while observing an ultrasound longitudinal image.
  Arms: ultrasound-guided caudal block

SUMMARY:
Surgical repair of the hip can be extremely painful and is associated with considerable postoperative pain in children despite the use of systemic opioids. These patients may benefit from neuraxial analgesia in adjunction with general anesthesia.

DETAILED DESCRIPTION:
Regional anesthetic techniques have been widely used for pain management in a variety of pediatric surgeries, as they increase the efficiency of postoperative pain control; minimize parenteral opioid requirements, and improve both patient and parent satisfaction as well. The erector spinae muscle plane block (ESB) is an evolving regional anesthetic technique gaining popularity in pediatric procedures. Erector spinae block is an effective regional anesthesia method as it blocks both somatic and visceral pain by injecting the local anesthetic solution into the inter-fascial space between the transverse process and the erector spinae muscle, it is performed by distributing local anesthetic into several paravertebral spaces. it was reported a successful ultrasound-guided ESP block performed at the L4 transverse process level provided postoperative analgesia in adult patients undergoing hip and proximal femur surgeries.

Caudal block (CB) is a well-established remarkable practice because of its simplicity, safety, and effectiveness. A single-shot caudal block with a local anesthetic agent, such as bupivacaine, is a standard procedure, and analgesia is provided during pediatric orthopedic surgeries in the lower limbs; unfortunately, its action stops early in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* • ASA I and II,

  * aged 2-7 years
  * scheduled for unilateral surgical hip reconstruction under general anaesthesia.

Exclusion Criteria:

* Children with spinal anomalies,

  * altered mental status or a history of developmental delay,
  * infection at the site of injection,
  * history of allergy to local anaesthetics
  * history of blood disease or coagulopathy,
  * Patient's guardian refusal to participate in the study

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry, Consolability (FLACC) Pain Scale 2 hours postoperative | first postoperative 24 hours
  To evaluate the quality of postoperative analgesia using the FLACC. Each category is scored on the 0-2 scale, which results in a total score of 0-10. 0=relaxed and comfortable, 1-3= mild discomfort, 4-6= moderate pain and 7-10= sever discomfort or pain or both

SECONDARY OUTCOMES:
time to the first analgesic request | recorded in hours for the first 24 hour
  the first time to pain scores are high and rescue analgesic is given
total analgesic requests | 24 hours
  total consumption of postoperative analgesics
Emergence agitation using Paediatric Anaesthesia Emergence Delirium (PAED) scale. | 24 hours
  PAED score ≥ 10 will be considered to be a diagnostic endpoint for the development of agitation. Emergence agitation and postoperative pain (scores of ≥ 10) will be managed by intravenous doses of fentanyl 0.5 mic/kg, repeated after 10 min if the child still agitated or in pain, with a maximum total dose of 2 mic/kg.

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa A Hassan, M.D., Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt